CLINICAL TRIAL: NCT06506032
Title: Clinical Effect and Wound Penetration of Vancomycin in Open-heart Surgery Patients Receiving Negative Pressure Wound Therapy for Deep Sternal Wound Infection
Brief Title: Vancomycin and Negative Pressure Therapy for Post-sternotomy Deep Sternal Wound Infection
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other); Masaryk University (Other); Masaryk Memorial Cancer Institute (Other); Technical University of Ostrava (Unknown)
Responsible Party: Sponsor
Other Study IDs: KCH-24-DSWI-vanko; 06/RVO-FNOs/2021 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2024-06-28; First posted 2024-07-17 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Post-Sternotomy Deep Sternal Wound Infection
Keywords: Exudate; Deep Sternal Wound Infection; Negative Pressure Wound Therapy; Open-Heart Surgery; Vancomycin; Wound Penetration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and exudate samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with NPWT with DSWI: Patients with deep sternal wound infection were enrolled in this study group.
  Interventions: Drug: Intravenous Vancomycin administration
- Patients without DSWI after cardiac surgery: Patients without deep sternal wound infection after cardiac surgery were enrolled in this study group.
  Interventions: Other: Standard postoperative therapy

INTERVENTIONS:
Drug: Intravenous Vancomycin administration — Vancomycin was administered to the patients at the discretion of the physician
  Groups: Patients treated with NPWT with DSWI
Other: Standard postoperative therapy — The patients received standard postoperative therapy
  Groups: Patients without DSWI after cardiac surgery

SUMMARY:
Only a limited number of studies have been published that monitored the penetration of antibiotics from blood into exudate in patients treated with negative pressure wound therapy (NPWT), and that evaluated the adequacy of current dosage regimens according to antibiotic tissue concentrations. A higher migration rate of several antibiotics (including vancomycin) to exudate has been reported in patients with skin ulcers, skin defects, burns, and traumatic wounds treated with NPWT compared to patients without NPWT.

In the present study, the investigators will evaluate the pharmacokinetic profile and wound penetration of vancomycin in open-heart surgery patients with post-sternotomy deep sternal wound infection receiving NPWT.

DETAILED DESCRIPTION:
For this prospective observational study, consecutive patients treated with NPWT for post-sternotomy deep sternal wound infection (DSWI) will be enrolled. On the first day of the study, serum and exudate samples will be synchronously collected at 0 (pre-dose), 0.5, 1, 2, 3, and 6 hours after vancomycin administration. On the following three consecutive days, additional samples will be collected, only before vancomycin administration.

The ratio of average vancomycin concentration in wound exudate to serum will be observed for free (unbound) and for total (bound + unbound) concentration. The percentage of free vancomycin in wound exudate and in serum will be observed. The level of vancomycin wound penetration will be observed for three days. The total hospital stay in patients with DSWI versus those without DSWI will be recorded, together with the in-hospital or 90-day mortality, together with late DSWI recurrence. All-cause mortality will be analyzed during a median follow-up of 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* clinical and laboratory signs of significant infection
* indication for NPWT with concomitant antibiotic therapy

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with deep sternal wound infection after open-heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Vancomycin penetration into exudate | repeated measurements for the total of 72 hours
  To determine the vancomycin penetration into the wound during NPWT, the investigators compared the vancomycin total (bound + unbound) average exudate concentration to the vancomycin total (bound + unbound) average serum concentration on the first study day. The same calculation was used to determine the penetration ratio for free (unbound) vancomycin concentrations on the first study day.
  For samples from three consecutive days, the investigators compared the vancomycin total (bound + unbound) through exudate concentrations with the vancomycin total (bound + unbound) through serum concentrations. The same calculation was used to determine the penetration ratio for free (unbound) vancomycin concentrations on three consecutive days.

SECONDARY OUTCOMES:
Identification of pre-, intra-, and postoperative risk factors for deep sternal wound infection (DSWI) development | 3 days
  The investigators will identify independent risk factors for DSWI by comparing patients with and without DSWI after cardiac surgery.
Recurrence of DSWI | 1- year follow-up
  The investigators will assess the recurrence of DSWI in the study subjects.
Determination of mortality | 1- year follow-up
  The investigators will assess the in-hospital, 90-day, and all-cause mortality in the study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kolek, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (5):
- Czechia (5):
  - University of Ostrava, Ostrava, Moravian-Silesian Region
  - Technical University of Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Masaryk University, Brno, South Moravian
  - Masaryk Memorial Cancer Institute, Brno, South Moravian

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Perezgrovas-Olaria R, Audisio K, Cancelli G, Rahouma M, Ibrahim M, Soletti GJ, Chadow D, Demetres M, Girardi LN, Gaudino M. Deep Sternal Wound Infection and Mortality in Cardiac Surgery: A Meta-analysis. Ann Thorac Surg. 2023 Jan;115(1):272-280. doi: 10.1016/j.athoracsur.2022.04.054. Epub 2022 May 23. PMID 35618048
- [Background] Baillot R, Cloutier D, Montalin L, Cote L, Lellouche F, Houde C, Gaudreau G, Voisine P. Impact of deep sternal wound infection management with vacuum-assisted closure therapy followed by sternal osteosynthesis: a 15-year review of 23,499 sternotomies. Eur J Cardiothorac Surg. 2010 Apr;37(4):880-7. doi: 10.1016/j.ejcts.2009.09.023. Epub 2009 Oct 31. PMID 19880326
- [Background] Polykandriotis E, Horch RE, Jost M, Arkudas A, Kees F, Schmitz M. Can systemically administered antibiotics be detected in wound tissues and surfaces under negative pressure wound therapy? Int Wound J. 2019 Apr;16(2):503-510. doi: 10.1111/iwj.13063. Epub 2019 Jan 3. PMID 30604928
- [Background] Ida Y, Matsumura H, Onishi M, Ono S, Imai R, Watanabe K. Measurement of vancomycin hydrochloride concentration in the exudate from wounds receiving negative pressure wound therapy: a pilot study. Int Wound J. 2016 Apr;13(2):204-8. doi: 10.1111/iwj.12260. Epub 2014 Mar 28. PMID 24674131
- [Background] Rowan MP, Niece KL, Rizzo JA, Akers KS. Wound Penetration of Cefazolin, Ciprofloxacin, Piperacillin, Tazobactam, and Vancomycin During Negative Pressure Wound Therapy. Adv Wound Care (New Rochelle). 2017 Feb 1;6(2):55-62. doi: 10.1089/wound.2016.0698. PMID 28224048
- [Derived] Kolek M, Duricova J, Brozmanova H, Sistik P, Jurica J, Kankova K, Motyka O, Kacirova I. Vancomycin wound penetration in open-heart surgery patients receiving negative pressure wound therapy for deep sternal wound infection. Ann Med. 2025 Dec;57(1):2444544. doi: 10.1080/07853890.2024.2444544. Epub 2024 Dec 23. PMID 39711425